CLINICAL TRIAL: NCT06482580
Title: Comparison of Effect of Ankle Exercise in PNF Pattern and Clam Exercise on Lower Extremity Muscle Strengh and Performance in Adults With Flexible Flat Feet: A Randomized Controlled Trial
Brief Title: The Effect of Different Exercises on Lower Extremity Performance in Flexible Flatfoot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Hande Esen, MSc, PT, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-77082166-604.01-930455
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Flexible Flatfoot
Keywords: Foot deformities; Intrinsic foot muscle training; Muscle strenghening; Short-foot exercises; Performance; Proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Flatfoot; Foot Deformities | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study was designed as an experimental, 3-arm parallel-group, double-blind randomized controlled trial with a 6-week intervention period.
  The study will be conducted at Toros University physiotherapy and exercise laboratory.
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary researcher will ensure blinding. Participants and the researcher conducting the assessments will be blinded to group information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNF exercise group (Experimental): All groups will be subjected to exercise training for 6 weeks: PNF exercise group will receive 3-dimensional (3D) foot-ankle extension exercise and short-foot exercise. The exercise will be performed 2 days a week under the supervision of a physiotherapist and 1 day as home exercise; KA exercise will be performed daily, 2 days under the supervision of a physiotherapist and the other days as home exercise.
  Interventions: Other: PNF exercise; Other: Short-foot exercise
- Clam exercise group (Experimental): All groups will be subjected to exercise training for 6 weeks: Clam exercise group will receive mussel exercise and short-foot exercise. The exercise will be performed 2 days a week under the supervision of a physiotherapist and 1 day as home exercise; KA exercise will be performed daily, 2 days under the supervision of a physiotherapist and the other days as home exercise.
  Interventions: Other: Clam exercise; Other: Short-foot exercise
- Control group (Active Comparator): All groups will be subjected to exercise training for 6 weeks: Control group will receive only KA exercise and this exercise will be performed daily, 2 days under the supervision of a physiotherapist and the other days as home exercise.
  Interventions: Other: Short-foot exercise

INTERVENTIONS:
Other: PNF exercise — Ankle and foot exercises practiced for 6 weeks.
  Arms: PNF exercise group
Other: Clam exercise — Hip exercise practiced for 6 weeks.
  Arms: Clam exercise group
Other: Short-foot exercise — Foot exercise practiced together for 6 weeks.

SUMMARY:
In the study, the effects of two different strengthening exercises combined with short foot exercise on lower extremity functional performance and muscle strength will be examined and compared in adults aged 18-45 years with flexible flatfoot. This study was designed as an experimental, 3-arm, parallel group, double-blind randomized controlled study that included a 6-week intervention period.

DETAILED DESCRIPTION:
Participants will be randomly divided into 3 different groups (control group, foot-ankle exercise group, hip exercise group). The control group will be instructed to perform only short foot exercise; the foot-ankle exercise group will be instructed to perform 3-dimensional foot-ankle extension exercise in proprioceptive neuromuscular facilitation (PNF) pattern in addition to short foot exercise; the hip exercise group will be instructed to perform hip abductor and external rotator muscle strengthening exercise (clam exercise) in addition to short foot exercise. Foot-ankle and hip exercises will be performed against resistance with the help of an elastic band, 3 days a week under the supervision of a physiotherapist and progression will be made by changing to a higher level of difficulty band color every 2 weeks. Short foot exercise will be performed every day of the week (3 days under the supervision of a physiotherapist; the rest of the days as a home exercise program) and will be progressed by changing position (sitting, standing, on one leg respectively) every 2 weeks. All exercises will be performed for 6 weeks. Assessments will be performed at the beginning and end of the exercises by another researcher blinded to group allocation. Isometric muscle strength of the intrinsic foot, four-way ankle circumference and hip abductor-external rotator muscles, endurance of the plantar flexors, forward jump and dynamic balance performance will be evaluated respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age range is 18-45 years
* Navicular drop is 10 mm or more
* Getting a value of +6 points or more from the Foot Posture Index-6

Exclusion Criteria:

* Orthopedic and rheumatological diseases of the spinal region and lower extremities
* Surgery history of the spine and lower extremities
* Neurological and systemic disorders
* Describe lower extremity and/or lower back pain in the last 6 months
* Disorders that may affect cognition and balance (otitis media, visual impairment, etc.)
* Body mass index being above normal values (18-24.9 kg/m2)
* Having rigid flat feet and/or hallux rigidus-limitus deformity
* Being involved in regular sports or exercise
* Having received any physiotherapy or rehabilitation treatment for flat feet or hips in the last year

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Medial longitudinal arch height | 6 weeks
  Medial longitudinal arch height will be evaluated with the navicular drop test.
Static foot posture | 6 weeks
  Static foot posture will be evaluated with Foot Posture Index-6.

SECONDARY OUTCOMES:
Isometric muscle strength | 6 weeks
  Abductor hallucis, flexor digitorum brevis, flexor hallucis brevis, 4-way ankle muscles and hip abductor/external rotator isometric muscle strength will be evaluated using a digital hand-held dynamometer.
Lower extremity functional performance | 6 weeks
  With plantar flexor focused endurance performance heel raise test; with dynamic balance Y balance test; Single leg forward jump performance will be evaluated with the single leg hop for distance test.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Esen, PhD. c, Principal Investigator — Gazi University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Gazi University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang C, Chen LY, Liao YH, Masodsai K, Lin YY. Effects of the Short-Foot Exercise on Foot Alignment and Muscle Hypertrophy in Flatfoot Individuals: A Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 22;19(19):11994. doi: 10.3390/ijerph191911994. PMID 36231295
- [Background] Engkananuwat P, Kanlayanaphotporn R. Gluteus medius muscle strengthening exercise effects on medial longitudinal arch height in individuals with flexible flatfoot: a randomized controlled trial. J Exerc Rehabil. 2023 Feb 23;19(1):57-66. doi: 10.12965/jer.2244572.286. eCollection 2023 Feb. PMID 36910682
- [Background] Okamura K, Fukuda K, Oki S, Ono T, Tanaka S, Kanai S. Effects of plantar intrinsic foot muscle strengthening exercise on static and dynamic foot kinematics: A pilot randomized controlled single-blind trial in individuals with pes planus. Gait Posture. 2020 Jan;75:40-45. doi: 10.1016/j.gaitpost.2019.09.030. Epub 2019 Sep 29. PMID 31590069
- [Background] Pabon-Carrasco M, Castro-Mendez A, Vilar-Palomo S, Jimenez-Cebrian AM, Garcia-Paya I, Palomo-Toucedo IC. Randomized Clinical Trial: The Effect of Exercise of the Intrinsic Muscle on Foot Pronation. Int J Environ Res Public Health. 2020 Jul 7;17(13):4882. doi: 10.3390/ijerph17134882. PMID 32645830